CLINICAL TRIAL: NCT01059292
Title: Department of Renal Transplantation, the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, China
Brief Title: TIPE2 Associated With Kidney Transplant
Acronym: TIPE2
Status: Suspended | Type: Observational
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Department of Renal Transplantation, the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an Jiaotong University
Other Study IDs: jia123456
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2009-10

CONDITIONS: Renal Transplant
Keywords: we have complieted party research

SUMMARY:
TIPE2, a negative regulator of innate and adaptive immunity that maintains immune homeostasis. The investigators want to know whether TIPE2 is a risk factor for graft loss and gives rise to the immune dysfunction in renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* long-term surival(>5year),AR and CR kidney transplant patients and healty Volunteers as control

Exclusion Criteria:

* without hepatitis , tumor and infections

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: kidney transplant patients and healty Volunteers
Sampling Method: Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2009-10